CLINICAL TRIAL: NCT05608980
Title: Effect of Hypochlorous Acid on Blepharitis Through Ultrasonic Atomization: a Randomized Clinical Trial
Brief Title: 0.01% Hypochlorous Acid in the Treatment of Blepharitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: ShuGuang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0.01% Hypochlorous Acid
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Blepharitis
Keywords: Blepharitis; Hypochlorous Acid; Eyelid cleanser; Eyelid hygiene; Meibomian gland dysfunction
MeSH Terms: conditions — Blepharitis; Meibomian Gland Dysfunction | interventions — Hypochlorous Acid

STUDY DESIGN:
Intervention Model Description: A prospective, controlled, randomized study.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Active Comparator): 0.01%hypochlorous acid group
  Interventions: Drug: 0.01% hypochlorous acid
- Placebo (Placebo Comparator): eyelid wipes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.01% hypochlorous acid — once daily 0.01% hypochlorous acid topical treatment via ultrasonic atomization for 2 weeks
  Other Names: 0.01%HOCI
  Arms: Treatment arm
Drug: Placebo — once daily eyelid wipes for 2 weeks
  Arms: Placebo

SUMMARY:
This is a multi-center, multidisciplinary, open-label, randomized controlled prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Anterior or mixed (anterior + posterior) blepharitis.
3. Similar clinical condition of both eyes.
4. A negative urine pregnancy test result for women of childbearing potential
5. Normal lid position and closure
6. Ability to understand and provide informed consent to participate in this study
7. Willingness to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

1. Any ocular surface disease other than blepharitis.
2. Known allergy to hypochlorous acid or boric acid.
3. Eye surgery in the last 6 months.
4. History of Stevens-Johnson syndrome or ocular pemphigoid
5. Ocular trauma in the last 6 months.
6. Use of contact lenses in the last 6 months.
7. Pregnancy or lactation.
8. Daily use of makeup on lashes.
9. Any ocular or systemic medication that might affect the ocular microbiota (antibiotics, immunosuppressants, steroids).
10. Pregnant or lactating women
11. Signs of current infection, including fever and current treatment with antibiotics
12. Liver, renal, or hematologic disease
13. The use of any other investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | Change from baseline OSDI at 2 weeks
  0-100 score based on the ocular surface disease index (OSDI) questionnaire
meibum quality | Change from baseline meibum quality score at 2 weeks
  Meibum quality were measured by using firm digital pressure applied over 5 lower lid glands. Meibum quality was graded as: grade 0, clear; grade 1, cloudy; grade 2, cloudy with granular debris; and grade 3, thick like toothpaste.
Corneal fluorescein staining | Change from baseline corneal fluorescein staining at 2 weeks
  scored by Oxford staining score
FBUT | Change from baseline FTBUT at 2 weeks
  fluorescent tear break up time fluorescein tear film break-up time

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxu Hong, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China